CLINICAL TRIAL: NCT03424746
Title: Pilot Trial of Limb Preservation Using Chelation Therapy in Diabetic Patients With Critical Limb Ischemia
Brief Title: Chelation Therapy in Diabetic Patients With Critical Limb Ischemia
Acronym: TACT-PAD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mt. Sinai Medical Center, Miami (Other)
Responsible Party: Principal Investigator, Gervasio Lamas, MD, Chair, Department of Medicine- Chief, Division of Cardiology, Mt. Sinai Medical Center, Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-36-H-07
Record Dates: First submitted 2018-01-31; First posted 2018-02-07 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Critical Limb Ischemia; Peripheral Arterial Disease
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease | interventions — Edetic Acid; Chelation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label EDTA chelation (Experimental): EDTA-based chelation therapy plus vitamins in diabetic patients with severe peripheral artery disease presenting with impending amputation and determine if there is an improvement in outcomes and a delay or reduction of amputations.
  Interventions: Drug: disodium EDTA

INTERVENTIONS:
Drug: disodium EDTA — Open-label study of TACT-formula, EDTA-based chelation therapy + commercially available TACT oral multi vitamins, delivering 40-50 infusions over 1 year.
  Other Names: chelation therapy

SUMMARY:
This is a Pilot Trial Using Chelation Therapy for Limb Preservation in Diabetic Patients with Critical Limb Ischemia.

DETAILED DESCRIPTION:
The purpose of this research study is to evaluate the effect of ethylenediaminetetraacetic acid (EDTA) based chelation therapy plus vitamins in diabetic patients with severe peripheral artery disease presenting with impending amputation and determine if there is an improvement in outcomes and a delay or reduction of amputations.

The investigators propose to enroll 10 patients in an open-label study of TACT-formula, EDTA-based chelation therapy + commercially available TACT oral multi vitamins, delivering 40-50 infusions over 1 year. Clinical assessment, and noninvasive blood flow assessments will be performed at baseline, and at completion of 20 and 40 infusions. HIPAA-compliant photographs of the affected lower limbs will be taken at each infusion visit.

The specific aims of this open-label pilot study are to:

1. Assess the effect of EDTA-based chelation therapy plus vitamins in diabetic patients with below-the-knee peripheral artery disease presenting with impending amputation and determine if there is an improvement in vascular flow parameters, such that the scheduled amputation can be averted or reduced in extent.
2. Co-primary severity endpoint: Changes in pain scores, quality of life, wound severity, segmental lower extremity pressures and endothelial function.
3. Assess safety of EDTA-based chelation therapy in this patient population, defined as deterioration of renal function, symptomatic hypocalcemia or hypoglycemia within 8 hours of each infusion, or Class 4 heart failure within 24 hours of an infusion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female older than 50 years of age;
* On treatment for diabetes mellitus, or fasting glucose 126 mg/dL or higher, or self-identified as diabetic
* Diagnostic of moderate or high-risk infra-popliteal chronic critical limb ischemia (Rutherford Clinical Severity Score 4 or 5) defined as:
* The presence of rest pain or non-healing ulceration for at least 2 weeks plus:
* A resting ankle systolic pressure (in either the dorsalis pedis or posterior tibial arteries) of ≤60 mmHg in the affected limb); or
* A resting toe systolic pressure of ≤40 mmHg in the affected limb or
* Skin perfusion pressure of ≤40 mmHg in the affected limb
* Significant stenosis (≥75%) of two or more infra-popliteal arteries in the affected limb as verified by one imaging technique (angiography, magnetic resonance angiography (MRA), computed tomographic angiography (CTA) or doppler examination) within 6 months prior to enrollment;
* Patients able to give informed consent.

Exclusion Criteria:

* Arterial insufficiency or ulcer in the lower extremity as the result of a non-atherosclerotic disorder.
* Subjects with evidence of active osteomyelitis or deep ulceration exposing bone or tendon in the extremity planned for treatment;
* Subjects in whom there is extensive heel ulceration
* Intravenous chelation therapy within 1 year (>5 infusions)
* Allergy to any study drug
* Symptomatic or clinically evident heart failure
* Heart failure hospitalization within 6 months
* Blood pressure >160/100
* No venous access
* Serum creatinine >2.0 mg/dL
* Platelet count <100000/mm3
* Cigarette smoking within the last 3 months
* Liver disease or Alanine aminotransferase (ALT), aspartate aminotransferase (AST) > 2.0 times the upper limit of normal
* Diseases of copper, iron, or calcium metabolism
* Inability to tolerate the study-required fluid load
* Inability to keep to study schedules
* Medical condition likely to affect patient survival within 4 years
* Women of child-bearing potential

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Improvement in vascular flow parameters | 1 year
  Segmental lower extremity pressures including Skin Perfusion Pressure (SPP), Pulse Volume Recording (PVR) and ankle brachial index (ABI), will be obtained at baseline, after 20 and 40 infusions using the SensiLase PAD-IQ® . This test can be used to accurately detect the presence and severity of peripheral artery disease. Additionally, for patients entering the continued treatment phase, the test will be performed during infusion visits 45 and 50.
Wound Evaluation | 1 Year
  HIPAA-compliant pictures of skin integrity including wounds and areas of gangrene will be obtained for each patient at baseline and every 5 infusions. Wound assessment includes ulcer measurements (length, width, depth and undermining) and percentage of epithelialization.
  Additionally, for patients entering the continued treatment phase, wound evaluation will be performed during infusion visits 45 and 50.
Peripheral Artery Questionnaire | 1 Year
  The severity of PAD will be assessed at baseline, 20th and 40th infusions, with a Peripheral Arterial Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gervasio Lamas, MD, Principal Investigator — Mount Sinai Medical Center of Florida
Locations (1):
- Mount Sinai Medical Center, Miami Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided